CLINICAL TRIAL: NCT01066767
Title: Randomized, 2-Way Crossover, Bioequivalence Study of Fexofenadine Hydrochloride 180 mg Tablets and Allegra® 180 mg Tablets Administered as 1 x 180 mg Tablet in Healthy Subjects Under Fed Conditions
Brief Title: Bioequivalence Study of Dr. Reddy's Laboratories Limited Fexofenadine Hydrochloride 180 mg Tablets Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Assistant Manager, Dr. Reddy's Laboratories Limited
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 02041
Record Dates: First submitted 2010-02-09; First posted 2010-02-10 (Estimated); Last update posted 2010-02-10 (Estimated); Status verified 2010-02

CONDITIONS: Healthy
MeSH Terms: interventions — fexofenadine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fexofenadine (Experimental): Fexofenadine Hydrochloride 180 mg Tablets Dr. Reddy's Laboratories Limited
  Interventions: Drug: Fexofenadine
- Allegra (Active Comparator): Allegra Tablets 180 mg Aventis Pharmaceuticals Inc.,
  Interventions: Drug: Fexofenadine

INTERVENTIONS:
Drug: Fexofenadine — Fexofenadine Hydrochloride 180 mg Tablets
  Other Names: Allegra 180 mg Tablets

SUMMARY:
Randomized, 2-Way Crossover, Bioequivalence Study of Fexofenadine Hydrochloride 180 mg Tablets of Dr.Reddy's Laboratories Limited, and Allegra® 180 mg Tablets aventis Administered as

1 x 180 mg Tablet in Healthy Subjects under Fed Conditions

DETAILED DESCRIPTION:
The objective of this study is to compare the rate and extent of absorption of fexofenadine hydrochloride 180 mg tablets (test) versus Allegra® (reference) administered as 1 x 180 mg tablet under fasting conditions. Single oral dose (1 x 180 mg) in each period with a washout of at least 7 days between doses.

ELIGIBILITY:
Inclusion Criteria:

Subjects enrolled in this study will be members of the community at large. The recruitment advertisements may be done using different media (e.g. radio, newspaper, Anapharm Inc.

Web site, Anapharm Inc. volunteers' data base). Subjects must meet all of the following criteria in order to be included in the study:

* Subjects will be females and/or males, smokers and non-smokers, 18 years of age and older.
* Female subjects will be post-menopausal or surgically sterilized.

  * Post-menopausal status is defined as absence of menses for the past 12 months or hysterectomy with bilateral oophorectomy at least 6 months ago.
  * Sterile status is defined as hysterectomy, bilateral oophorectomy or tubal ligation at least 6 months ago.

Exclusion Criteria:

* Subjects to whom any of the following applies will be excluded from the study:

  * Clinically significant illnesses within 4 weeks of the administration of study medication.
  * Clinically significant surgery within 4 weeks prior to the administration of the study medication.
  * Any clinically significant abnormality found during medical screening.
  * Any reason which, in the opinion of the medical sub investigator, would prevent the subject from participating in the study.
  * Abnormal laboratory tests judged clinically significant.
  * Positive urine drug screen at screening.
  * Positive testing for hepatitis B, hepatitis C or HN at screening.
  * ECG abnormalities (clinically significant) or vital sign abnormalities (systolic blood pressure lower than 90 or over 140 mmHg, or diastolic blood pressure lower than 50 or over 90; or heart rate less than 50 bpm or over 100 bpm) at screening.
  * Subjects with BMl ≥ 30.0.
  * History of significant alcohol abuse within six months of the screening visit or any indication of the regular use of more than two units of alcohol per day (1 Unit = 150 mL of wine or 360 mL of beer or 45 mL of alcohol 40%).
  * History of drug abuse or use of illegal drugs: use of soft drugs (such as marijuana) within 3 months of the screening visit or hard drugs (such as cocaine, phencyclidine (PCP) and crack) within 1 year of the screening visit.
  * Any food allergy, intolerance, restriction or special diet that, in the opinion of the medical Sub investigator, contraindicates the subject's participation in this study.
  * History of allergic reactions to fexofenadine hydrochloride or its ingredients.
  * History of allergic reactions to heparin.
  * Use of any drugs known to induce or inhibit hepatic drug metabolism (examples of inducers: barbiturates, carbamazepine, phenytoin, glucocorticoids, rifampin/rifabutin; examples of inhibitors: antidepressants, cimetidine, diltiazem, erythromycin, ketoconazole, MAO inhibitors, neuroleptics, verapamil, quinidine), use of an investigational drug or participation in an investigational study within 30 days prior to administration of the study medication.
  * Use of prescription medication within 14 days prior to administration of study medication or over-the-counter products (including natural products, vitamins, garlic as supplement)within 7 days prior to administration of study medication, except for topical products without systemic absorption.
  * Subjects who have a depot injection or an implant of any drug 3 months prior to administration of study medication.
  * Donation of plasma (500 mL) within 7 days. Donation or loss of whole blood prior to administration of the study medication as follows:
  * less than 300 mL of whole blood within 30 days or
  * 300 mL to 500 mL of whole blood within 45 days or
  * more than 500 mL of whole blood within 56 days.
  * Smoking more than 25 cigarettes per day.

Additional exclusion criteria for females only:

* Breast-feeding subjects.
* Positive urine pregnancy test at screening (performed on all females).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2002-04; Primary Completion 2002-05 (Actual); Study Completion 2002-05 (Actual)

PRIMARY OUTCOMES:
Bioequivalence study of Dr. Reddys, Fexofenadine Hydrochloride 180 mg tablets | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Girard, M.D, Principal Investigator — Anapharm
Locations (1):
- Anapharm Inc.,, Sainte-Foy Quebec, Canada